CLINICAL TRIAL: NCT01605747
Title: A Blinded Placebo Controlled Clinical Outcomes Study of Culturelle® in the Prophylaxis of Infection and Diarrhea
Brief Title: Study of Culturelle in the Prophylaxis of Infection and Diarrhea
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was stopped due to inavailability of subjects meeting eligibility criteria.
Sponsor: Shriners Hospitals for Children (Other)
Responsible Party: Principal Investigator, Michele Gottschlich, Director, Nutrition Services, Shriners Hospitals for Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 10-12-13-02
Record Dates: First submitted 2012-05-08; First posted 2012-05-25 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Pediatric Burns

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Culturelle (Experimental)
  Interventions: Dietary Supplement: Culturelle
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Culturelle — one capsule 2x per day per feeding tube
  Arms: Culturelle
Dietary Supplement: Placebo — one placebo 2x per day per feeding tube
  Arms: Placebo

SUMMARY:
The primary objective of this study is to determine if probiotic prophylaxis has immunologic and gastrointestinal advantages in pediatric burn patients.

ELIGIBILITY:
Inclusion Criteria:

* acute burn injury
* consented within 10 days of injury
* feeding tube present-

Exclusion Criteria:

* GI disorder prior to burn
* milk allergy or insensitivity
* non-burned

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2013-01 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Infectious outcome | 3 years
  Record incidence of infection between the experimental and placebo groups.

SECONDARY OUTCOMES:
Clinical outcome | 3 years
  Plan to measure clinical outcome between the experimental and placebo groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Shriners Hospital for Children, Cincinnati, Ohio, United States